CLINICAL TRIAL: NCT04890938
Title: Sputum-guided Treatment With Comprehensive Care Management for Respiratory Improvement to Provide Value and Escalate Care - A Randomized-controlled Trial
Brief Title: Sputum-guided Treatment With Comprehensive Care Management in COPD - A Randomized-controlled Trial
Acronym: STRIVE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: McMaster University (Other)
Collaborators: Hamilton Academic Health Sciences Organization (Other); St. Joseph's Healthcare Hamilton (Other); Hamilton Health Sciences Corporation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 13532
Record Dates: First submitted 2021-05-13; First posted 2021-05-18 (Actual); Last update posted 2024-11-21 (Actual); Status verified 2024-11

CONDITIONS: COPD
Keywords: COPD; Exacerbation; Comprehensive care management; Sputum
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Who Masked: Care Provider
Masking Description: Study personnel (aside from the research coordinator) will be blinded to randomization, sputum biomarker results, and treatment arm. Sputum biomarker results (de-identified) will be available to site leads to optimize treatment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sputum-guided management and comprehensive care management (Experimental): The intervention consists of 6-months of CCM and sputum biomarker-directed treatment of airway inflammation, including hospital and clinic visits. Clinic visits at 2, 6, and 16 weeks. The key elements of CCM will be provided, including case management, self-management education, and coordination of community/hospital resources (1). Clinic nurse will review inhaler technique with the patient. Sputum (spontaneous) biomarkers will be measured with results used to direct therapy at the time of AECOPD and during clinic visits after hospital discharge, at both sites.
  Interventions: Combination Product: Sputum-guided management and comprehensive care management
- Usual Care (Active Comparator): This group will also receive clinic visits at 2, 6, and 16 weeks with a study physician, and also education material, inhaler technique assessment and education, and case management from the clinic personnel. The study physician will pursue further investigation and/or further intervention if they see fit.
  Interventions: Other: Usual Care

INTERVENTIONS:
Combination Product: Sputum-guided management and comprehensive care management — Those in the intervention group will have their treatment determined by the presence and type of airway inflammation whether during AECOPD or as part of clinic optimization. Corticosteroids are given for airway eosinophilia (sputum eosinophils >3%), and antibiotics for airway neutrophilia (sputum neutrophils ≥65% and total cells >10 million cells/gram) or a positive sputum culture. Specialized stains to identify aspiration (Oil Red O; (3)) and left ventricular dysfunction (Perl's Prussian blue; (4)) will guide swallowing assessment and cardiac work-up, respectively. If a sputum sample is not produced as an outpatient spontaneously, then sputum induction will be pursued 8 weeks after discharge. If there are no sputum samples to guide inhaler regimen, then it will be determined by the study physician guided by the Canadian Thoracic Society guidelines (2) if a sputum-guided regimen has not already been established.
  Arms: Sputum-guided management and comprehensive care management
Other: Usual Care — As per previous, this group will receive three follow-up visits with study pulmonologist and clinic personnel interventions.
  Arms: Usual Care

SUMMARY:
Chronic obstructive pulmonary disease (COPD) is a lung condition affecting 1 in 6 Canadians and does not have a cure. Flare-ups of COPD are the most common reason someone goes to hospital in Canada. This is made worse because within 30-days of having a flare-up, 1 in 5 patients will come back to hospital for the same problem.

Flare-ups of COPD often have many causes and these are different person to person. Sometimes it is related to behaviours such as smoking or not using medicines properly. Other times, it is from lung inflammation. Education programs that help people learn about their disease and maintain healthy behaviours, and using phlegm to decide on which medicines will be useful, have been studied separately and appear to work, but many people still have flare-ups. To help fix this problem, we need to look carefully at each patient, to make sure they are on the right medicine but also have the right behaviours and support to benefit from medical care.

The goal of this project is to see if patients who are taught the right behaviours and have their lung inflammation controlled with the right medicines will have fewer COPD flare-ups than those who get normal care.

DETAILED DESCRIPTION:
STRIVE is a randomized-controlled trial comparing a two-pronged intervention, including sputum-biomarker-directed treatment of airway inflammation, and comprehensive care management, to usual care, for COPD patients with frequent exacerbation from two sites.

The intervention consists of 6-months of comprehensive care management (CCM) and sputum biomarker-directed treatment of airway inflammation, including hospital and clinic visits. Clinic visits will occur at 2, 6 and 16 weeks after hospital discharge. For the intervention group, the key elements of CCM will be provided, including case management, self-management education, and coordination of community/hospital resources (1). Spontaneous sputum biomarkers will be used to direct therapy at the time of AECOPD and during clinic visits after hospital discharge.

ELIGIBILITY:
Inclusion Criteria:

* >=2 exacerbations of COPD in the last 12-months, FEV1/FVC<0.7 or radiologic emphysema, with a >-10 pack-year smoking history

Exclusion Criteria:

* severe mental illness not controlled by medication or life-expectancy less than 6-months

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 128 (Estimated)
Dates: Start 2022-05-27 (Actual); Primary Completion 2025-03 (Estimated); Study Completion 2025-08 (Estimated)

PRIMARY OUTCOMES:
Severe exacerbations of COPD | 6 months
  As defined by an acute worsening of respiratory symptoms requiring treatment with antibiotics or steroids associated with ER visit or hospitalization.

SECONDARY OUTCOMES:
Moderate COPD Exacerbation | 6 months
  as defined by worsening of symptoms requiring the use of antibiotics or steroids without ER visit or hospitalization
Mild COPD Exacerbation | 6 months
  Defined as worsening of symptoms that were self-managed and resolved without systemic steroids or antibiotics; captured by Clinical COPD Questionnaire
COPD exacerbation associated with inflammation | 6 months
  Defined as an exacerbation (as defined previously) with an abnormal sputum cell count or sputum culture
Time to first COPD exacerbation associated with inflammation | 6 months
  Defined as time to an exacerbation (as defined previously) with an abnormal sputum cell count or sputum culture
Time to first COPD exacerbation | 6 months
  Defined as time to an exacerbation (as defined previously)
Change in Clinical COPD Questionnaire | 26 weeks
  Change in Clinical COPD Questionnaire between Week 0 and Week 26.
Change in COPD Assessment Test | 26 weeks
  Change in COPD Assessment Test between Week 0 and Week 26.
Change in Patient Health Questionnaire-9 | 26 weeks
  Change in Patient Health Questionnaire-9 between Week 0 and Week 26.
Change in General Anxiety Disorder-7 questionnaire | 26 weeks
  Change in General Anxiety Disorder-7 questionnaire between Week 0 and Week 26.
EQ-5D-5L questionnaire | 26 weeks
  Change in EQ-5D-5L between Week 0 and Week 26.
FEV1 | 16 weeks
  Change in FEV1 between clinic visits 1 and 3.
Sputum eosinophil percentage | 16 weeks
  Change in sputum eosinophil percentage between clinic visits 1 and 3
Sputum neutrophil count | 16 weeks
  Change in sputum neutrophil count between clinic visits 1 and 3
Sputum abnormalities rectified | 16 weeks
  The number of subjects who have their sputum abnormalities rectified will be recorded between clinics 1 and 3
Use of oral or inhaled corticosteroid | 6 months
  Cumulative dose of oral and inhaled corticosteroid
Use of antibiotics | 6 months
  Cumulative courses of oral or intravenous antibiotics
Participant recruitment number | 2 years
  number of patients approached for recruitment during study
Reason for non-participation | 2 years
  reasons for non-participation during recruitment period
Clinic attendance | 6 months
  Number of clinic visits attended while enrolled in the study
Number of days to visit 1 | Should fall within a 2-3 week window
  number of days to visit 1 from hospital discharge
Number of clinic visits | 6 months
  Number of clinic visits patients attend during the 6 months that they are participating in the study
Patient care | study duration
  number of nursing telephone calls initiated by the patient, number of adequate sputum samples collected, and the number referred to a smoking cessation program
Side effects | 26 weeks
  Side effects will be captured by noting peak serum glucose levels and blood pressure measured in-hospital, and the occurrence of psychosis, candidiasis, C. difficile infection, and gastrointestinal upset as reported by the patient during clinic visits

CONTACTS AND LOCATIONS:
Overall Officials: Terence Ho, MB, MSc, Principal Investigator — St. Joseph's Healthcare Hamilton
Locations (2):
- Canada (2):
  - Hamilton General Hospital, Hamilton, Ontario
  - St. Joseph's Healthcare Hamilton, Hamilton, Ontario

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Nici L, ZuWallack R. Integrated Care in Chronic Obstructive Pulmonary Disease and Rehabilitation. COPD. 2018 Jun;15(3):223-230. doi: 10.1080/15412555.2018.1501671. Epub 2018 Sep 5. PMID 30183417
- [Background] Bourbeau J, Bhutani M, Hernandez P, Marciniuk DD, Aaron SD, Balter M, et al. CTS position statement: Pharmacotherapy in patients with COPD-An update. Canadian Journal of Respiratory, Critical Care, and Sleep Medicine. 2017;1(4):222-41.
- [Background] Wilson AM, Nair P, Hargreave FE, Efthimiadis AE, Anvari M, Allen CJ; ELVIS Research Study Group. Lipid and smoker's inclusions in sputum macrophages in patients with airway diseases. Respir Med. 2011 Nov;105(11):1691-5. doi: 10.1016/j.rmed.2011.07.011. Epub 2011 Aug 9. PMID 21831624
- [Background] Leigh R, Sharon RF, Efthimiadis A, Hargreave FE, Kitching AD. Diagnosis of left-ventricular dysfunction from induced sputum examination. Lancet. 1999 Sep 4;354(9181):833-4. doi: 10.1016/S0140-6736(99)80018-X. PMID 10485730